CLINICAL TRIAL: NCT03271112
Title: Frailty Prevention in Elderly People From Reunion Island: Effects of Adaptated Exercises on Physical Performance
Brief Title: Frailty Prevention in Elders From Reunion Island
Acronym: 5P-PILOTE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Collaborators: Centre National de la Recherche Scientifique, France (Other); Institut de Recherche pour le Developpement (Other Government); General Social Security Fund (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2017/CHU/00
Record Dates: First submitted 2017-08-31; First posted 2017-09-01 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Frail Elderly Syndrome; Physical Activity
MeSH Terms: conditions — Motor Activity | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: Pilote study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise program (Other): Participation to the 12-wks exercise program
  Interventions: Other: Exercise program

INTERVENTIONS:
Other: Exercise program — Measurement of physical performance before and after the 12 wks-exercice program

SUMMARY:
In Reunion Island, people encounter environmental and social conditions leading to premature ageing and subsequent frailty. Social welfare has developped exercise programs to promote physical activity especially for elderly with higher risk factors of frailty, including low incomes.

The study evaluates the potent benefit effect of such exercise program on physical performance and frailty improvement in seniors from Reunion Island. All seniors participate to a 12-weeks exercise program especially dedicated to this targeted population needs and ability.

DETAILED DESCRIPTION:
Regular physical activity has been shown to slow down sarcopenia, and increase strengh in elders. Nevertheless, senior with low incomes do not usually have access to physical activity areas.

Social partners are in close relationship with these elders and could promote free exercise programs dedicated to elders classified as "GIR5-6" according to the French scale "AGIRR". The AGIRR scale takes into account several criteria allowing the evaluation of the level of autonomy. The level of autonomy is closely related to frailty and could be reversed since elders have not reach a dependant-state. The "GIR5-6" level means that elderly people are still not dependant but exhibit several frailty risk factors.

The level of frailty and the physical performance of the participants is assessed by standard geriatric evaluation before the 12-wks exercice program. The improvement of the physical performance is assessed after he 12-wks exercice program.

ELIGIBILITY:
Inclusion Criteria:

* Retired
* with an autonomy level corresponding to the "GIR 5-6" level of the French "AGIRR scale"
* informed consent

Exclusion Criteria:

* physical activity prohibited
* under guardianship

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2017-09-04 (Actual); Primary Completion 2019-05-07 (Actual); Study Completion 2019-07-04 (Actual)

PRIMARY OUTCOMES:
Physical performance improvement | Physical performance improvement from baseline to 12 wks
  Physical performance is assessed as as balance, walk and strength improvement

SECONDARY OUTCOMES:
Quality of life score | SF36 improvement from baseline to 12 wks
  Improvement of quality of life assessed by SF36 v1 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marc EYCHENE, MD, Principal Investigator — Centre Hpospitalier Universitaire de La REUNION
Locations (1):
- Chu Reunion Island, Saint-Joseph, Reunion

IPD SHARING:
Plan to Share IPD: No